CLINICAL TRIAL: NCT04295590
Title: Impact of Augmenting Exercise Intensity vs. Frequency on Peak Work Rate
Brief Title: Impact of Augmenting Exercise Intensity vs. Frequency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brendon Gurd, PhD (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor-Investigator, Brendon Gurd, PhD, Professor, School of Kinesiology & Health Studies, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UCD Study
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Exercise Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frequency then Intensity (Experimental): Training period 1: Frequency comparison Training period 2: Intensity comparison
  Interventions: Behavioral: Frequency comparison; Behavioral: Intensity comparison
- Intensity then Frequency (Experimental): Training period 1: Intensity comparison Training period 2: Frequency comparison
  Interventions: Behavioral: Frequency comparison; Behavioral: Intensity comparison

INTERVENTIONS:
Behavioral: Frequency comparison — One leg assigned to low-frequency low-intensity (3 days per week of 11 x 1 min @ 73% peak work rate interspersed with 1-minute periods of active recovery). The other leg assigned to high-frequency low-intensity (5 days per week of 11 x 1 min @ 73% peak work rate interspersed with 1-minute periods of active recovery).
Behavioral: Intensity comparison — One leg assigned to low-frequency low-intensity (3 days per week of 11 x 1 min @ 73% peak work rate interspersed with 1-minute periods of active recovery). The other leg assigned to low-frequency high-intensity (3 days per week of 8 x 1 min @ 100% peak work rate interspersed with 1-minute periods of active recovery).

SUMMARY:
The purpose of this study is to compare the impact of augmenting exercise intensity and augmenting exercise frequency on peak work rate. Participants will complete exercise tests and provide 8 skeletal muscle samples following a within-subjects randomized crossover design utilizing single-leg cycling. Both training periods will be 4 weeks long and skeletal muscle biopsies will be collected from both legs before and after each training period. All exercise sessions will be supervised, take place in the investigator's laboratory, and occur on stationary bikes.

ELIGIBILITY:
Inclusion Criteria:

* Recreational active (<3 hours per week of aerobic exercise)
* Willing to provide skeletal muscle biopsies

Exclusion Criteria:

* Cardiovascular or metabolic disease
* Athletes or individuals exceeding 3 hours per week of aerobic exercise
* Smokers

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
Peak work rate | Before exercise training on two days (~7 and 6 days before first training session; ~24 hours apart), and after exercise on two days (~48-96 hours after the last training session; ~24 hours apart)
  Change in Highest work rate achieved (30s period) during incremental exercise tests

SECONDARY OUTCOMES:
Peak oxygen uptake | Before exercise training on two days (~7 and 6 days before first training session; ~24 hours apart), and after exercise on two days (~48-96 hours after the last training session; ~24 hours apart)
  Change in Highest oxygen uptake achieved (30s period) during incremental exercise tests
Maximal citrate synthase activity | Before exercise training (~7 days before first training session), and after exercise training (~48-72 hours after the last training session)
  Change in maximal citrate synthase activity

CONTACTS AND LOCATIONS:
Overall Officials: Brendon J Gurd, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's Muscle Physiology Lab in the School of Kinesiology and Health Studies at Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No